CLINICAL TRIAL: NCT01761201
Title: "A Prospective, Randomized, Comparative Clinical Trial of the Efficacy and Safety of Levofloxacin Versus Isoniazid in the Treatment of Latent Tuberculosis Infection in Liver Transplant Patients".
Brief Title: "Efficacy and Safety of Levofloxacin vs Isoniazid in Latent Tuberculosis Infection in Liver Transplant Patients".
Acronym: FLISH-ILT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment rythm not sufficent to reach the simple size needed.
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Network for Research in Infectious Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLISH-ILT; 2010-022302-41 (EudraCT Number)
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Latent Tuberculosis Infection; Infection in Solid Organ Transplant Recipients
Keywords: Prophylaxis; Tuberculosis; Transplant recipients; Transplant waiting list
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — Levofloxacin; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- levofloxacin (Experimental): Levofloxacin 500 mg daily for 9 months starting on the waiting list for liver transplant
  Interventions: Drug: Levofloxacin
- Isoniazid (Active Comparator): Isoniazid 300 mg/day for 9 months beginning after transplantation, when the "liver function is stable" and not before 3 months nor after 6 months
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin
  Other Names: Generic name: Levofloxacin; ATC Code: J01MA.; Pharmaceutical form: Levofloxacin 500 mg film-coated tablets
  Arms: levofloxacin
Drug: Isoniazid — 300 mg/day for 9 months beginning after transplantation, when the "liver function is stable" and not before 3 months nor after 6 months.
  Other Names: Generic name: Isoniazid.; ATC Code: J04AC; Pharmaceutical form: tablets.
  Arms: Isoniazid

SUMMARY:
A multicenter, prospective, non-inferiority, randomized and open clinical trial comparing levofloxacin with isoniazid in the treatment of latent tuberculosis infection in patients eligible for liver transplantation.

Patients over 18 years of age on the waiting list for liver transplantation.

Sample size: n=870 patients.

HYPOTHESIS

Levofloxacin treatment of latent tuberculosis infection, begun while on the waiting list for liver transplantation, is safer and not less effective than isoniazid treatment begun after transplantation when liver function is stable.

DETAILED DESCRIPTION:
Primary Objective

1. To demonstrate that the incidence of tuberculosis in patients with latent tuberculosis infection and treated with levofloxacin is not higher than that observed in patients treated with isoniazid.

   Secondary Objective
2. To demonstrate that the efficacy of levofloxacin is not limited by adverse effects, paying particular attention to hepatotoxicity.

ELIGIBILITY:
Inclusion Criteria:

Liver transplantation candidates with age ≥ 18 years, no clinical or radiological evidence of active tuberculosis and negative pregnancy test (if applicable)who must meet one or more of the following criteria:

* PPD skin test (initial or after a "booster effect") >5 mm. Alternatively, the determination may be made by the interferon gamma (IFN-g) production in PPD-stimulated lymphocytes using the Quantiferon-TB or ELISPOT assays.
* Past history of tuberculosis not properly treated.
* Past history of contact with a patient with active TB.
* Chest x-ray consistent with past untreated TB (apical fibronodular lesions, calcified solitary nodule, calcified lymph nodes or pleural thickening).

The patient must give their written informed consent.

Exclusion Criteria:

* Lack of consent to participate in the study.
* Intolerance or allergy to levofloxacin or to isoniazid.
* Documented contact with tuberculosis resistant to levofloxacin or to isoniazid.
* Treatment in the previous month with drugs with potential activity against Mycobacterium tuberculosis, (especially quinolones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Difference in incidence of tuberculosis disease | 18 months of follow-up
  A patient will be considered as having tuberculosis when Mycobacterium tuberculosis is isolated by culture or M. Tuberculosis DNA is isolated from a representative clinical sample, organ fluid or tissue by polymerase chain reaction. Also cases of histopathologically confirmed tuberculosis (caseating granulomas with/without demonstration of acid-alcohol resistant bacillus [BAAR]) and clinically compatible presentation will be accepted. Tuberculosis will be classified as pulmonary (pulmonary parenchymal involvement), extrapulmonary (involvement of different organs to the lung) or disseminated (involvement of at least two non-contiguous organs). Cases where tuberculosis is diagnosed on the basis of clinical and/or radiology suspicion and for whom the corresponding physician has prescribed a specific treatment will not be accepted.

SECONDARY OUTCOMES:
Mortality | 18 months
  Number of deaths of any cause
Toxicity | During all the 18 months of follow-up
  Occurrence of grade 3 or 4 toxicities according to the grading (severity) scale of the National Cancer Institute Common Toxicity Criteria Version 4.0, NCI-CTC-AE v 4.0.
Retransplantation | 18 months
  A new liver transplantation during the follow-up
Graft dysfunction | 18 months
  Development of advanced graft fibrosis stages 3 and 4
Transplant rejection | 18 months
  The occurrence of acute rejection or chronic rejection as per conventional definitions during the follow-up.

OTHER OUTCOMES:
Safety | 18 months
  Drug tolerance will be evaluated by a clinical study interview and periodic analytical determinations which will include levels of transaminases (ALT and AST), alkaline phosphatase and gamma-GT, bilirubin, according to the study visit schedule.
  All symptoms and laboratory results will be evaluated for severity according to the grading (severity) scale of the National Cancer Institute Common Toxicity Criteria Version 3.0, NCI-CTC-AE v 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Julián de la Torre Cisneros, MD, Principal Investigator — Hospital Universitario Reina Sofía, Córdoba, Spain; José M. Aguado, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre, Madrid
Locations (18):
- Spain (18):
  - Complejo Hospitalario Universitario, A Coruña
  - Complejo Hospitalario de Albacete, Albacete
  - Hospital Infanta Cristina,, Badajoz
  - Hospital Clinic, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Reina Sofía, Córdoba
  - Hospital universitario Virgen de las Nieves, Granada
  - Hospital 12 de Octubre, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Marqués de Valdecillas, Santander
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Background] Torre-Cisneros J, Doblas A, Aguado JM, San Juan R, Blanes M, Montejo M, Cervera C, Len O, Carratala J, Cisneros JM, Bou G, Munoz P, Ramos A, Gurgui M, Borrell N, Fortun J, Moreno A, Gavalda J; Spanish Network for Research in Infectious Diseases. Tuberculosis after solid-organ transplant: incidence, risk factors, and clinical characteristics in the RESITRA (Spanish Network of Infection in Transplantation) cohort. Clin Infect Dis. 2009 Jun 15;48(12):1657-65. doi: 10.1086/599035. PMID 19445585
- [Background] Aguado JM, Herrero JA, Gavalda J, Torre-Cisneros J, Blanes M, Rufi G, Moreno A, Gurgui M, Hayek M, Lumbreras C, Cantarell C. Clinical presentation and outcome of tuberculosis in kidney, liver, and heart transplant recipients in Spain. Spanish Transplantation Infection Study Group, GESITRA. Transplantation. 1997 May 15;63(9):1278-86. doi: 10.1097/00007890-199705150-00015. PMID 9158022
- See also: official web site for the Spanish Infectious Disease Network — http://www.reipi.org/index.php/es/